CLINICAL TRIAL: NCT05172921
Title: The Role of Environmental Factors in Thyroid Cancer
Brief Title: Environmental Factors and Thyroid Cancer
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Maaike A Van Gerwen, Assistant Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-21-01547
Record Dates: First submitted 2021-12-23; First posted 2021-12-29 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — Dried blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Exposed: High exposure to environmental pollutants
- Non-exposed: Low exposure to environmental pollutants

SUMMARY:
Thyroid cancer incidence has been steadily increasing and has nearly tripled since the 1970's in the US and worldwide. Early detection of small, papillary thyroid cancers using high quality diagnostic imaging explains only about 50% of this increased incidence, suggesting that there is a true increase in the occurrence of thyroid cancer and that changes in the prevalence of environmental risk factors might play a role in thyroid cancer etiology and progression. Yet, the cascade of environmental triggers linked to thyroid cancer remains elusive.

'Exposomics' studies all health relevant chemical exposures that an individual experiences, and leverages metabolomic platforms to estimate the "internal" environment, informing both exogenous exposures and the metabolic products that lead to, or arise from, disease. Besides exposure to ionizing radiation as known modifiable risk factor, epidemiological evidence suggests that exposure to endocrine disrupting chemicals may be a potential thyroid cancer risk factor due to their known effects on thyroid function. However, these studies relied either on exposure questionnaires which are susceptible to recall bias, or used a limited set of targeted biomarkers measured after diagnosis for testing associations with case-control status, and not thyroid cancer prognosis. Further, the molecular basis for observed associations with thyroid cancer remains unclear.

To address the overall hypothesis that environmental exposures alter metabolic pathways and therefore affect thyroid cancer prognosis, small amounts of blood will be collected using dried blood microsampler technology (e.g. Mitra® sampling devices), which is minimally invasive and can be used to collect repeated blood measurements at home, without the need for specialized training. These dried blood samples will be used to perform metabolomics experiments, which describe the sum of exogenous exposures, metabolic alterations, and biological response. Additional exposure assessment will be performed using an exposure questionnaire. These results will be associated with thyroid cancer prognosis, e.g. disease-specific survival, disease recurrence, and mutational profiles, thus investigating the role of environmental exposures in the development of more aggressive forms of thyroid cancer.

ELIGIBILITY:
Inclusion criteria:

* Bethesda category III, IV, V or VI following Fine Needle Aspiration; if a patient has a benign tumor following surgery, patient data/ samples will be stored to serve as benign control in potential future projects.
* Age 18 years and older
* Surgical candidate
* Ability to provide informed consent

Exclusion criteria:

* History of thyroid cancer
* Completion surgery candidate
* Pregnant women or other vulnerable patients (e.g. wards of the state, prisoners)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thyroid cancer patients seen within the Mount Sinai Health System
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2035-09 (Estimated)

PRIMARY OUTCOMES:
Phospholipids | 4 years
  Using Liquid Chromatography-High Resolution MS (LC-HRMS) analysis, exposure profiles will be ascertain for existing of combination(s) of plasma metabolites (endogenous and exogenous) that act synergistically to increase risk of non-familial, papillary thyroid cancer.
  Phospholipids is an endogenous metabolite
Ceramides | 4 years
  Using Liquid Chromatography-High Resolution MS (LC-HRMS) analysis, exposure profiles will be ascertain for existing of combination(s) of plasma metabolites (endogenous and exogenous) that act synergistically to increase risk of non-familial, papillary thyroid cancer.
  Ceramides is an endogenous metabolite
per-and polyfluoroalkyl substances (PFAS) | 4 years
  Using Liquid Chromatography-High Resolution MS (LC-HRMS) analysis, exposure profiles will be ascertain for existing of combination(s) of plasma metabolites (endogenous and exogenous) that act synergistically to increase risk of non-familial, papillary thyroid cancer.
  per-and polyfluoroalkyl substances (PFAS) is an exogenous metabolite

CONTACTS AND LOCATIONS:
Overall Officials: Maaike van Gerwen, MD, PhD, Principal Investigator — MSH
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to make IPD available to other researchers. Researchers will have access to the data/ samples in a de-identified manner.